CLINICAL TRIAL: NCT04359862
Title: Sedation With Sevoflurane Versus Propofol in Patients With Acute Respiratory Distress Syndrome Caused by COVID19 Infection
Acronym: SEVO-COVID19
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low recruitment ratio
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SEVO-COVID19
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Acute Respiratory Distress Syndrome; COVID19 Infection
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19 | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Intervention Model Description: Multicenter, national, randomized, 1:1 ratio, controlled, parallel, open study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SEVOFLURANE Group (Experimental)
  Interventions: Drug: Sevoflurane
- PROPOFOL Group (Active Comparator)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane — 25 patients sedated with Sevoflurane via inhalation, starting with 6 ml/h and changing every 15 minutes until an adequate level of sedation is achieved ( BIS 40-50)
  Arms: SEVOFLURANE Group
Drug: Propofol — 25 patients standard sedation with intravenous propofol, starting with 2 mg/kg/h and changing every 15 minutes until an adequate level of sedation is achieved ( BIS 40-50)
  Arms: PROPOFOL Group

SUMMARY:
It is a multicenter, national, randomized 1:1 ratio, controlled, parallel, open study.

Patients with severe ARDS-CoVid19 will be included in the trial within the first 24 hours.

Patients will be randomized to one of the treatment groups:

* SEV group: 25 patients with Sevoflurane sedation by inhalation, starting at 6 ml/h and changing every 15 minutes until an adequate level of sedation is achieved (BIS 40-50)
* PRO group: 25 patients standard sedation with intravenous propofol, starting with 2 mg/kg/h and changing every 15 minutes until an adequate level of sedation is achieved ( BIS 40-50)

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or more.
* Diagnosis of Acute Respiratory Distress Syndrome caused by COVID19 infection.
* Signature of Patient's Consent or Verbal Consent of Legal Representative

Exclusion Criteria:

* Intracranial hypertension
* Hypersensitivity to the active ingredient (propofol or sevoflurane) or to any of the excipients
* Current volume < 250ml
* History of malignant hyperthermia
* Liver failure
* Neutropenia (<0.5x109)
* Pregnant or lactating women
* Have received chemotherapy in the last month since their inclusion in the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
PaO2/FiO2 | Day 2
  To evaluate the effect of 48-hour treatment with inhaled sevoflurane on arterial oxygenation, assessed by PaO2/FiO2 on day two, in patients with ARDS-CoVid19

SECONDARY OUTCOMES:
TNFα | Day 2
  To quantify the effects of sevoflurane on pro-inflammatory cytokine levels during ARDS-CoVid19
IL-1b | Day 2
  To quantify the effects of sevoflurane on pro-inflammatory cytokine levels during ARDS-CoVid19
IL-6 | Day 2
  To quantify the effects of sevoflurane on pro-inflammatory cytokine levels during ARDS-CoVid19
IL-8 | Day 2
  To quantify the effects of sevoflurane on pro-inflammatory cytokine levels during ARDS-CoVid19
Mortality | Day 30
  To evaluate the 30-day mortality.

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospital Universitario Cruces, Barakaldo, Bizkaia
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No